CLINICAL TRIAL: NCT03269201
Title: Mapping Functional Networks of Brain Activity (Brain Network Activation, BNA) Based on Analysis of Evoked Response Potential (ERP) EEG Signals in Patients With Movement Disorders
Brief Title: Brain Network Activation in Patients With Movement Disorders
Acronym: BNA-MDi
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Sharon Hassin, Director, Movement Disorders Institute., Sheba Medical Center
Other Study IDs: 4408-17
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia; Normal Pressure Hydrocephalus; Cerebellar Ataxia; Multiple System Atrophy; Progressive Supranuclear Palsy; Corticobasal Degeneration; Dementia With Lewy Bodies
Keywords: parkinsonism; ataxia; tremor; dystonia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Hydrocephalus, Normal Pressure; Cerebellar Ataxia; Multiple System Atrophy; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Lewy Body Disease; Parkinsonian Disorders; Ataxia; Tremor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Parkinson;s Disease: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.
- Essential tremor: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis.Additionally patients will be rated using mmse/ MoCA, Verbal Fluency, essential tremor rating assessment scale (TETRAS) clinical rating scale for tremor (CRST).SF-EMG and KinesiaOne and motion sensor assessment writing and drawing on digitizer, for tremor.
- Multiple system atrophy: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.
- Normal Pressure Hydrocephalus: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - TIMED UP AND GO TASK (INSTRUMENTAL)
- DYSTONIA-focal, generalized and others: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.Fahn-Marsden Evaluation Scale for Dystonia
  .SF-EMG and KinesiaOne and motion sensor assessment , writing and drawing on digitizer,for dystonia
- Cerebellar ataxia: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency,Scale for the assessment and rating of ataxia (SARA), International Cooperative Ataxia Rating Scale . TIMED UP AND GO TASK (INSTRUMENTAL)
- Progressive supranuclear palsy: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.
- Corticobasal degeneration: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.
- Dementia with Lewy Bodies: Patients will undergo EEG recordings at rest and while performing the set of motor and cognitive tasks and BNA analysis. Additionally patients will be rated using MoCA, FAB, Verbal Fluency, - Beck Depression Inventory, PDQ-39, PD sleep scale (PDSS), MDS-UPDRS.SF-EMG and KinesiaOne and motion sensor assessment for tremor.

SUMMARY:
The diagnosis and management of movement disorders, such as Parkinson's disease (PD), parkinson-plus syndromes (PPS), dystonia, essential tremor (ET), normal pressure hydrocephalus (NPH) and others is challenging given the lack of objective diagnostic and monitoring tools with high sensitivity and specificity. A cornerstone in research of neurological disorders manifesting as MDi is the investigation of neurophysiological changes as potential biomarkers that could help in diagnosis, monitoring disease progression and response to therapies. Such a neuro-marker that would overcome the major disadvantages of clinical questionnaires and rating scales (such as the Unified Parkinson's disease rating scale -UPDRS, for PD, The Essential Tremor Rating Assessment Scale -TETRAS, for ET and others), including low test-retest repeatability and subjective judgment of different raters, would have real impact on disease diagnosis and choice of interventions and monitoring of effects of novel therapeutics, including disease modifying therapies.

To address this, ElMindA has developed over the last decade a non-invasive, low-cost technology named Brain Network Activation (BNA), which is a new imaging approach that can detect changes in brain activity and functional connectivity. Results from proof-of concept studies on PD patients have demonstrated that: 1) PD patients exhibited a significant decrease in BNA scores relatively to healthy controls; 2) notable changes in functional network activity in correlation with different dopamine-agonist doses; 3) significant correlation between BNA score and the UPDRS). 4) BNA could also differentiate early PD from healthy controls

DETAILED DESCRIPTION:
Objective: The primary aim of the current project is to assess the utility of the BNA as a quantitative, objective, neurophysiological marker for diagnosis and monitoring of the above most common MDi in man.

The secondary aim is to find predictive bio-types (electrophysiological fingerprint) of the above MDi and within these disorders identifying patients with high likelihood of developing: 1) psychiatric complications such as dopaminergic medication induced-impulse control disorder (ICD) for PD; 2) Depression; 3) Gait and balance Impairment; or 4) Cognitive deterioration, including (PD-MCI) or PD-dementia (PDD).

The technology: BNA technology is based on non-invasive recordings of multi-channel EEG event-related potentials (ERPs), and a comprehensive multi-dimensional analysis of such recordings, aimed at understanding and visualizing the network complexity (or Brain Networks Activation patterns) of brain function. BNA takes cognitive ERPs, a direct measure of neural activity associated with cognitive functions, to a new frontier, unparalleled by EEG, QEEG or ERP alone or by any other anatomic and functional brain imaging and evaluation tools. The BNA algorithms use innovative sets of signal processing, pattern recognition and machine learning techniques to seek and map activated neural pathways while patients are engaged in a cognitive task. The resulting BNA network patterns can aid clinicians with profiling of changes in functionality and/or dysfunctionality. BNA received an FDA clearance and a CE mark approval during 2014, and is commercially available in the US, with more than 20 active clinical and research sites focusing on numerous neurological and neuropsychological disorders. More than 30,000 data sets of functional brain networks of healthy subjects have been already collected and may serve as normative data for comparison.

ELIGIBILITY:
Inclusion Criteria:

* For PD: Idiopathic PD patients (according to the UK PD Society brain bank clinical diagnostic criteria (bradykinesia plus at least one other cardinal feature of PD, no atypical features or secondary cause).
* For ET: bilateral, largely symmetrical postural or kinetic tremor involving hand and forearms that is visible and persistent. Additional or isolated tremor of the head may occur but in the absence of abnormal posturing.
* For Parkinson plus syndrome: multiple system atrophy (MSA), progressive supranuclear palsy (PSP), corticobasal degeneration (CBD) and dementia with Lewy bodies (DLB).
* For NPH: patients exhibiting some or all components of the clinical triad consisting of gait disturbance, urinary control disturbance and cognitive impairment as well as proof of enlarged ventricular system or hydrocephalus by cranial CT or MRI scans.
* For Dystonia: patients exhibiting a movement disorder syndrome in which sustained or repetitive muscle contractions result in twisting and repetitive movements or abnormal fixed postures. The movements may resemble a tremor. Patients included will be those with either idiopathic, toxic or hereditary mechanism.
* For Cerebellar ataxia: patients exhibiting impairment of coordination and balance as part of an ataxic cerebellar syndrome which is caused by degeneration of the cerebellum and its afferent and efferent connections due to various etiologies, such as genetic or sporadic neurodegenerative processes or others.

Exclusion Criteria:

* In the investigator's opinion, any unstable or clinically significant condition that would impair the participants' ability to comply with study requirements.
* Patients with significant psychiatric symptoms or history or treatment with neuroleptics.
* MMSE <10
* Currently with lice or open wounds on scalp.
* Significant sensory deficits, e.g., deafness or blindness
* Current drug abuse or alcoholism.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 300 patients with MDs:
  Idiopathic PD , ET, PPS, NPH, dystonia and CAs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS part III score | 3 years
  Motor severity

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale | 3 years
  scale for ataxia
TETRAS | 3 years
  The Essential Tremor Rating Assessment Scale (TETRAS)
MDS-UPDRS total score | 3 years
  General measure for PD
MoCA Montreal - Cognitive Assessment | 3 years
  Cognitive Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Clinic, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Reches A, Nir RR, Shram MJ, Dickman D, Laufer I, Shani-Hershkovich R, Stern Y, Weiss M, Yarnitsky D, Geva AB. A novel electroencephalography-based tool for objective assessment of network dynamics activated by nociceptive stimuli. Eur J Pain. 2016 Feb;20(2):250-62. doi: 10.1002/ejp.716. Epub 2015 May 11. PMID 25960035
- [Background] Reches A, Levy-Cooperman N, Laufer I, Shani-Hershkovitch R, Ziv K, Kerem D, Gal N, Stern Y, Cukierman G, Romach MK, Sellers EM, Geva AB. Brain Network Activation (BNA) reveals scopolamine-induced impairment of visual working memory. J Mol Neurosci. 2014 Sep;54(1):59-70. doi: 10.1007/s12031-014-0250-6. Epub 2014 Feb 18. PMID 24535560
- [Background] Reches A, Laufer I, Ziv K, Cukierman G, McEvoy K, Ettinger M, Knight RT, Gazzaley A, Geva AB. Network dynamics predict improvement in working memory performance following donepezil administration in healthy young adults. Neuroimage. 2014 Mar;88:228-41. doi: 10.1016/j.neuroimage.2013.11.020. Epub 2013 Nov 21. PMID 24269569
- [Background] Sang L, Zhang J, Wang L, Zhang J, Zhang Y, Li P, Wang J, Qiu M. Alteration of Brain Functional Networks in Early-Stage Parkinson's Disease: A Resting-State fMRI Study. PLoS One. 2015 Oct 30;10(10):e0141815. doi: 10.1371/journal.pone.0141815. eCollection 2015. PMID 26517128
- [Background] Gao LL, Wu T. The study of brain functional connectivity in Parkinson's disease. Transl Neurodegener. 2016 Oct 28;5:18. doi: 10.1186/s40035-016-0066-0. eCollection 2016. PMID 27800157